CLINICAL TRIAL: NCT05448183
Title: A Single-arm, Open-label, Multi-center Phase II Clinical Study to Evaluate the Safety and Efficacy of Toripalimab Injection Combined With TACE in the Treatment of Extrahepatic Cholangiocarcinoma
Brief Title: An Observational Real World Study on the Efficacy and Safety of Toripalimab Injection Combined With TACE in the Treatment of Extrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuhua Duan (Other)
Responsible Party: Sponsor-Investigator, Xuhua Duan, Associate chief physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiECRCT20220189
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Extrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — toripalimab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab combined withTACE (Experimental)
  Interventions: Drug: Toripalimab, Gemcitabine,Oxaliplatin

INTERVENTIONS:
Drug: Toripalimab, Gemcitabine,Oxaliplatin — Toripalimab, 240mg, IV infusion, every 3 weeks (q3w), combined withTACE (Gemcitabine 1000mg/m2 , Oxaliplatin 135mg/m2) in a cycle of 3 weeks(q3w).

SUMMARY:
This is an open-label, single-arm, multicenter phase II clinical study to preliminarily observe and evaluate the efficacy and safety of Toripalimab combined with TACE in the treatment of extrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 75 years
* both men and women
* ECOG performance status score 0-2 points
* Child-Pugh score ≤ 7 points
* Expected survival ≥ 12 weeks
* Patients with histologically or cytologically confirmed extrahepatic cholangiocarcinoma, patients with obstructive jaundice need to return to normal after drainage
* At least one measurable lesion [spiral CT scan ≥ 10 mm (CT scan slice thickness no greater than 5 mm)] (RECIST Version 1.1)
* Vital organ function meets the following requirements: a. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; b. Platelets ≥ 75 × 109/L; c. Hemoglobin ≥ 8 g/dL; d. Serum albumin ≥ 2.8 g/dL; e. Bilirubin ≤ 3 ULN, ALT/AST ≤ 2.5 UILN; if there is liver metastasis, ALT/AST ≤ 5 times ULN; f. Creatinine clearance ≥ 50 mL/min (Cockcroft-Gault, see Appendix III); g. Normal thyroid function. h. Adequate cardiac function, 2-dimensional cardiac ultrasound examination of the score (LVEF) > 50%
* No history of serious drug allergy
* Women of childbearing age must have taken reliable contraceptive measures or have a pregnancy test before enrollment
* The subject voluntarily participates in this study. Sign the informed consent form, with good compliance and cooperation in follow-up

Exclusion Criteria:

* Known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs and their components
* Presence of any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; complete remission of asthma in childhood, no intervention after adulthood can be included; patients with asthma requiring bronchodilators for medical intervention can not be included)
* Patients are using immunosuppressive agents, or systemic hormone therapy to achieve the purpose of immunosuppression (dose > 10 mg/day prednisone or other effective hormones), and continue to use 2 times before enrollment
* Pregnant or lactating women
* Other malignant tumors have been diagnosed within 5 years before the first use of the study drug, except for effectively treated cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma and/or effectively resected in situ cervical cancer and/or breast cancer
* Patients prone to infection and poor blood glucose control
* Incomplete important imaging examination and incomplete record of adverse reactions
* Previous surgery, chemotherapy, targeted, radiotherapy and immune-related therapy
* Other conditions that the investigator judges may affect the conduct of the clinical study and the judgment of the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 1 year
  PFS is defined as time from the start of treatment to progression of disease or death.

SECONDARY OUTCOMES:
Objective response rate | Up to 1 year
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
Disease control rate | Up to 1 year
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.

CONTACTS AND LOCATIONS:
Overall Officials: Hua xu Duan, Doctor, Study Director — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Hennan, China

IPD SHARING:
Plan to Share IPD: Undecided